CLINICAL TRIAL: NCT05970003
Title: Comparative Effects of Copenhagen and Holmich Exercises in Hip Adductor Related Groin Pain, Strength and Lower Extremity Function in Soccer Players
Brief Title: Comparative Effects of Copenhagen and Holmich Exercises in Hip Adductor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR & AHS/23/0412
Record Dates: First submitted 2023-06-27; First posted 2023-08-01 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Groin Strain
Keywords: Holmich protocol; Copenhagen exercises; groin pain; adductor strain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Copenhagen exercise (Active Comparator): Group A will receive the Copenhagen exercise, also known as the adductor strengthening protocol, is a dynamic and high-intensity exercise. It doesn't require any special equipment and can be done in any training center.
  There are 3 different levels of exercise were performed by players.
  1. Level 1: Side-lying hip adduction exercise.
  2. Level 2: Copenhagen adduction exercises while both arms support at the knee.
  3. Level 3: Copenhagen adduction exercise - primary support at the ankle and minor support at the knee.
  Interventions: Other: Copenhagen exercises
- Group B : Holmich Exercises (Active Comparator): Group B will receive Holmich continues to provide the strongest evidence for the efficacy of exercise as an ARGP treatment.
  The Holmich treatment protocol exercise includes static and dynamic and/or isometric and isotonic strengthening exercises for hip adductors and abductors and also for abdominal muscles.
  There are 6 Different types of exercises were performed by players who were a participant with 3 sets of 10 repetitions with 15 sec recovery period.
  Interventions: Other: Holmich exercises

INTERVENTIONS:
Other: Copenhagen exercises — Group A performs copenhagen exercises
  Both groups will perform their routine warm ups and cool downs the total duration of the protocol is 6 weeks, 3 times a week the duration of each session 3 sets of 10 repetitions with 15 sec recovery period. Hip extensor and flexor stretching and strengthening.
  Arms: Group A: Copenhagen exercise
Other: Holmich exercises — The Holmich treatment protocol exercise includes static and dynamic and/or isometric and isotonic strengthening exercises for hip adductors and abductors and also for abdominal muscles.
  There are 6 Different types of exercises were performed by players who were a participant with 3 sets of 10 repetitions with 15 sec recovery period.
  Both groups will perform their routine warm ups and cool downs the total duration of the protocol is 6 weeks, 3 times a week the duration of each session 3 sets of 10 repetitions with 15 sec recovery period. Hip extensor and flexor stretching and strengthening.
  Arms: Group B : Holmich Exercises

SUMMARY:
Groin pain that relates to the adductor muscle usually represents in the groin region specifically in superior internal thigh. Tears or strains may happen within the muscles itself, tears or strains mainly occurs at musculotendinous junctions or within the tendons. Adductor strain is a familiar but mostly ignored cause of groin injury and pain among athletes. Risk factors include past hip or groin injury, age, weak adductors, muscle fatigue, lessen range of motion, and deficient stretching of the adductor muscle complex.

DETAILED DESCRIPTION:
This study will be a randomized clinical trial and will be conducted in Pakistan sports board and coaching center. Non-probability consecutive sampling will be used to collect the data. Sample size of this research is 46 subjects with age group between 18-30 years will be taken. Data will be collected from the patients of adductor strain that causes groin pain by using tools Numeric Pain Rating Scale for pain, Adductor Muscle Strength Test by Hand Held Dynamometer, The Copenhagen Hip and Groin Outcome Score (HAGO's) questionnaire and Lower Extremity Functional Scale (LEFS). An informed consent will be taken. Squeeze test will be performed to evaluate the adductor related groin pain. The subjects will be divided into two groups i.e. Group A and Group B. Group A will receive the Copenhagen exercise, also known as the adductor strengthening protocol, is a dynamic and high-intensity exercise. It doesn't require any special equipment and can be done in any training center. Group B will receive Holmich continues to provide the strongest evidence for the efficacy of exercise as an ARGP treatment. Both groups will perform their routine warm ups and cool downs the total duration of the protocol is 6 weeks, 3 times a week the duration of each session 3 sets of 10 repetitions with 15 sec recovery period Keywords groin pain, Holmich protocol, Copenhagen exercise, adductor strain.

ELIGIBILITY:
Inclusion Criteria:

* • Male soccer player age group 18-30 years

  * Groin pain during or after game
  * Persistent groin pain over 2-3 weeks
  * Pain at palpation of groin
  * Positive pain with Adductor squeeze test

Exclusion Criteria:

* • Low back pain

  * Infection (UTI)
  * Malignancy
  * Recent fractures or injuries
  * Hip osteoarthritis
  * Inguinal hernia

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 46 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Numerical pain rating scale (NPRS) | upto 4th weeks
  Numeric Pain Rating Scale for Pain In a Numerical Rating Scale (NRS), patients are asked to circle the number between 0 and 10, 0 and 20 or 0 and 100 that fits best to their pain intensity. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible.
Lower Extremity Functional Scale (LEFS) | upto 4th weeks
  Lower Extremity Functional Scale (LEFS) The Lower Extremity Functional Scale (LEFS) is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. The LEFS can be used by clinicians as a measure of patients' initial function, ongoing progress and outcome, as well as to set functional goals. The LEFS can be used to evaluate the functional impairment of a patient with a disorder of one or both lower extremities. It can be used to monitor the patient over time and to evaluate the effectiveness of an intervention.
  The final version of the LEFS consists 20 items, each with a maximum score of 4. The total possible score of 80 indicates a high functional level (Appendix). The scale is one page, can be filled out by most patients in less than 2 minutes, and is scored by tallying the responses for all of the items. Scoring is performed without the use of a calculator or computer and requires approximately 20 seconds
Manual Muscle Testing | upto 4th weeks
  MMT grades are usually labelled with the following terms: "zero," "trace," "poor," "fair," "good," and "normal." In addition, manual muscle testing grades can be further described using a numerical scale from 0 through 5.

CONTACTS AND LOCATIONS:
Overall Officials: Samrood Akram, Mphil, Principal Investigator — Riphah International University,Lahore
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mercurio M, Corona K, Galasso O, Cerciello S, Morris BJ, Guerra G, Gasparini G. Soccer players show the highest seasonal groin pain prevalence and the longest time loss from sport among 500 athletes from major team sports. Knee Surg Sports Traumatol Arthrosc. 2022 Jun;30(6):2149-2157. doi: 10.1007/s00167-022-06924-5. Epub 2022 Mar 8. PMID 35258646
- [Background] Haroy J, Clarsen B, Wiger EG, Oyen MG, Serner A, Thorborg K, Holmich P, Andersen TE, Bahr R. The Adductor Strengthening Programme prevents groin problems among male football players: a cluster-randomised controlled trial. Br J Sports Med. 2019 Feb;53(3):150-157. doi: 10.1136/bjsports-2017-098937. Epub 2018 Jun 10. PMID 29891614
- [Background] Schaber M, Guiser Z, Brauer L, Jackson R, Banyasz J, Miletti R, Hassen-Miller A. The Neuromuscular Effects of the Copenhagen Adductor Exercise: A Systematic Review. Int J Sports Phys Ther. 2021 Oct 1;16(5):1210-1221. doi: 10.26603/001c.27975. eCollection 2021. PMID 34631242
- [Background] Almeida MO, Silva BN, Andriolo RB, Atallah AN, Peccin MS. Conservative interventions for treating exercise-related musculotendinous, ligamentous and osseous groin pain. Cochrane Database Syst Rev. 2013 Jun 6;2013(6):CD009565. doi: 10.1002/14651858.CD009565.pub2. PMID 23740671